CLINICAL TRIAL: NCT02901574
Title: Cerebellar Transcranial Direct Current Stimulation to Augment Chronic Aphasia Treatment
Brief Title: Cerebellar Transcranial Direct Current Stimulation and Aphasia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00100024; R00DC015554 (NIH)
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- tDCS plus computerized naming therapy (Active Comparator): Anodal or cathodal tDCS, 2 milliamps (mA) plus computerized naming treatment for 15 sessions (20 minutes per each 45 minute treatment session) over the course of 3-5 weeks.The electrical current will be administered to the right cerebellum. The stimulation will be delivered at an intensity of 2 mA for a maximum of 20 minutes. Language therapy will be a computer delivered naming +picture matching task.
  Interventions: Device: Anodal or Cathodal tDCS; Behavioral: Computerized naming therapy
- Sham plus computerized naming therapy (Sham Comparator): Sham tDCS plus computerized naming treatment for 15 sessions (20 minutes per each 45 minute treatment session) over the course of 3-5 weeks. Current will be administered in the in a ramp like fashion for 15-30 seconds but then the current is gradually decreased and drop to 0 mA. Language therapy will be a computer delivered naming +picture matching task.
  Interventions: Device: Sham; Behavioral: Computerized naming therapy

INTERVENTIONS:
Device: Anodal or Cathodal tDCS — 2 mA or Anodal or Cathodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge (anode in group anode or cathode in group cathode) is placed on the right cerebellum. The stimulation will be delivered at an intensity of 2 mA in a ramp-like fashion for a maximum of 20 minutes.
  Arms: tDCS plus computerized naming therapy
Device: Sham — 2 mA of Anodal tDCS or Cathodal tDCS is induced between two 5cm X 5cn saline soaked sponges where one sponge (anode in group Anode and cathode in group Cathode) is placed on the right cerebellum. Ramping up of the current to 2 mA occurs over 15-30 seconds to allow participants to habituate to the tingling sensation. Then, the current will be ramped back down to 0 mA in the sham condition. Termination of the stimulation after the ramping up process is generally undetectable, and the brief duration of stimulation yields no functional effects.
  Arms: Sham plus computerized naming therapy
Behavioral: Computerized naming therapy — Computer delivered naming treatment requires matching (heard and seen being produced by the speaker) with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red button if the word does not match the picture.

SUMMARY:
People with post-stroke aphasia are left with some degree of chronic deficit for which current rehabilitative treatments are variably effective. This study investigates the behavioral and neural effects of multiple consecutive cerebellar tDCS sessions coupled with computerized naming therapy in stroke survivors with aphasia.

DETAILED DESCRIPTION:
The investigators will study the effect of right cerebellar transcranial direct current stimulation (tDCS) stimulation during language therapy for naming in individuals with chronic aphasia (>6 months post stroke). Naming difficulties are a persistent and common symptom in aphasia after left-hemisphere (LH) stroke. Although the interventions to improve naming can have benefits, a massive number of treatment sessions is usually required to show gains, particularly in individuals with chronic, large LH stroke. tDCS is a promising adjunct to traditional language therapy. tDCS is a safe, non-invasive, non-painful electrical stimulation of the brain which modulates cortical excitability by application of weak electrical currents in the form of direct current brain polarization. It is usually administered via saline-soaked surface sponge electrodes attached to the scalp and connected to a direct current stimulator with low intensities. Prior investigators have mainly focused on the role of LH in language recovery, wherein the electrode is placed in the left frontal or temporal region. However, in individuals with large lesions involving key language areas like the frontal and temporal cortex, it may be difficult to find viable tissue to stimulate in the LH. This study uses a novel electrode placement for chronic stroke patients with aphasia with large LH lesions. Targeting the intact right cerebellum allows for the possibility of identifying a single target that can be used across groups of people with aphasia with varying lesion sites and size in the LH. Evidence from functional neuroimaging and clinical studies indicate that the right cerebellum is important for both language and cognitive functions.

The investigators will utilize a randomized, double-blind, sham controlled, within-subject crossover trial design. A random subset (half) of participants will be assigned to the "anode" group (Group Anode) and other half will be assigned to the 'cathode' group (Group Cathode). Participants will take part in 2 intervention periods of 15 computerized naming training sessions (3-5 sessions per week), with either tDCS + naming therapy or sham+ naming therapy, separated by 2 months. Detailed language evaluation will take place before, immediately after, 2 weeks and 2 months post-intervention for each condition. The investigators will test the hypothesis that anodal tDCS or cathodal tDCS over the cerebellum and computerized naming therapy is associated with greater gains in accuracy in naming pictures, compared to sham combined with the same computerized naming therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have sustained a left hemisphere stroke.
* Participants must be fluent speakers of English by self-report.
* Participants must be capable of giving informed consent or indicating another to provide informed consent.
* Participants must be age 18 or older.
* Participants must be premorbidly right handed.
* Participants must be at least 6 months post stroke.
* Participants must have an aphasia diagnosis as confirmed by the Boston Diagnostic Aphasia Examination (BDAE) Short Form.
* Participants must achieve at least 65% accuracy on screening task (comparable to treatment task) on 1 of 3 attempts

Exclusion Criteria:

* Participants with lesion involving the right cerebellum
* Previous neurological or psychiatric disease.
* Seizures during the previous 12 months.
* Uncorrected visual loss or hearing loss by self-report.
* Use of medications that lower the seizure threshold (e.g., methylphenidate, amphetamine salts).
* Use of N-methyl-D-aspartate receptor (NMDA) antagonists (e.g., memantine).
* > 80% (140 out of 175) correct responses on the Philadelphia Naming Test at baseline.
* History of brain surgery or any metal in the head.
* Scalp sensitivity (per participant report).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajani Sebastian, PhD, CCC-SLP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the projects and dissemination of primary study results, the analysis data files will be made available to the public, along with the final version of the study protocol, the data dictionary, and brief instructions ("read me" file). The public use data files and the accompanying documents will be made available through the National Technical Information Service (NTIS).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants who were randomized did not start the intervention due to the COVID-19 pandemic and 1 did not start due to transportation issues.
Groups:
- tDCS Plus Computerized Naming Therapy First, Then Sham Plus Computerized Naming Therapy: Anodal or cathodal tDCS, 2 milliamps (mA) plus computerized naming treatment for 15 sessions (20 minutes per each 45 minute treatment session) over the course of 3-5 weeks.The electrical current will be administered to the right cerebellum. The stimulation will be delivered at an intensity of 2 mA for a maximum of 20 minutes. Language therapy will be a computer delivered naming +picture matching task.
  Anodal or Cathodal tDCS: 2 mA or Anodal or Cathodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge (anode in group anode or cathode in group cathode) is placed on the right cerebellum. The stimulation will be delivered at an intensity of 2 mA in a ramp-like fashion for a maximum of 20 minutes.
  Computerized naming therapy: Computer delivered naming treatment requires matching (heard and seen being produced by the speaker) with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red button if the word does not match the picture.
  Participants switch to the Sham plus computerized naming therapy after this.
- Sham Plus Computerized Naming Therapy First, Then tDCS Plus Computerized Naming Therapy: Sham tDCS plus computerized naming treatment for 15 sessions (20 minutes per each 45-minute treatment session) over the course of 3-5 weeks. Current will be administered in a ramp like fashion for 15-30 seconds but then the current is gradually decreased and drop to 0 mA. Language therapy will be a computer delivered naming +picture matching task.
  Sham: 2 mA of Anodal or Cathodal tDCS is induced between two 5cm X 5cm saline soaked sponges where one sponge (anode in group Anode and cathode in group Cathode) is placed on the right cerebellum. Ramping up of the current to 2 mA occurs over 15-30 seconds and then the current will be ramped back down to 0 mA in the sham condition. Termination of the stimulation after the ramping up process is generally undetectable, and the brief duration of stimulation yields no functional effects.
  Computerized naming therapy: Computer delivered naming treatment requires matching with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red button if the word does not match the picture.
  Participants then switch to tDCS plus computerized naming therapy after this.
Period: Intervention Period 1 (up to 5 Weeks)
Arm/Group | tDCS Plus Computerized Naming Therapy First, Then Sham Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy First, Then tDCS Plus Computerized Naming Therapy
Started | 14 | 14
Completed | 11 | 13
Not Completed | 3 | 1
Period: Wash Out ( 8 Weeks)
Arm/Group | tDCS Plus Computerized Naming Therapy First, Then Sham Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy First, Then tDCS Plus Computerized Naming Therapy
Started | 11 | 13
Completed | 10 | 12
Not Completed | 1 | 1
Period: Intervention Period 2 (up to 5 Weeks)
Arm/Group | tDCS Plus Computerized Naming Therapy First, Then Sham Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy First, Then tDCS Plus Computerized Naming Therapy
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants in this study meant to receive both of the interventions (tDCS and sham) in this cross-over design
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.71 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
Boston Diagnostic Aphasia Examination Aphasia Severity Rating Scale [Mean (Full Range); unit: units on a scale] — The scale ranges from 0-5. A score of 0 indicates no usable speech or auditory comprehension. A score of 5 indicates minimal discernible speech handicap.
  units on a scale | 2.71 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Change in Accuracy of Naming Untrained Pictures (Philadelphia Naming Test:PNT) Pre-treatment to Post-treatment
Description: To determine whether tDCS coupled with computerized naming therapy will improve naming performance of participants with post stroke aphasia more effectively than naming therapy alone (i.e., the sham condition).The PNT is a 175-item picture naming test where a person earns one point per each correct answer. Scores range from 0-175 with higher scores associated with better performance.
Time Frame: Before and after 15 sessions (3-5 sessions per week; up to 5 weeks) of treatment.
Population: Completers sample. Missing data is not imputed. Data was missing for 3 participants for tDCS and 1 participant for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Sham Plus Computerized Naming Therapy: Sham tDCS plus computerized naming treatment for 15 sessions (20 minutes per each 45 minute treatment session) over the course of 3-5 weeks. Current will be administered in the in a ramp like fashion for 15-30 seconds but then the current is gradually decreased and drop to 0 mA. Language therapy will be a computer delivered naming +picture matching task.
  Sham: 2 mA of Anodal tDCS or Cathodal tDCS is induced between two 5cm X 5cn saline soaked sponges where one sponge (anode in group Anode and cathode in group Cathode) is placed on the right cerebellum. Ramping up of the current to 2 mA occurs over 15-30 seconds, then, the current will be ramped back down to 0 mA in the sham condition. Termination of the stimulation after the ramping up process is generally undetectable, and the brief duration of stimulation yields no functional effects.
  Computerized naming therapy: Computer delivered naming treatment requires matching (heard and seen being produced by the speaker) with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red button if the word does not match the picture.
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 23 | 23
score on a scale | 5.76 [1.20 to 10.32] | 1.88 [-1.95 to 5.72]
Statistical Analysis 1: Comparison: tDCS Plus Computerized Naming Therapy vs Sham Plus Computerized Naming Therapy; Test type: Superiority; p = 0.24, Mixed Models Analysis — Threshold for significance is two-sided alpha of 0.05; Mean Difference (Final Values) = 3.87, 95% CI 2-sided [-2.55 to 10.30]

2. Secondary Outcome: Change in Accuracy of Naming Untrained Pictures (Philadelphia Naming Test:PNT)Pre-treatment to 2 Weeks Post-treatment.
Description: as for outcome 1
Time Frame: Pre-treatment and at 2 weeks Post-treatment
Population: Completers sample. Missing data is not imputed. Data was missing for 5 participants for the tDCS and 4 participants for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Sham Plus Computerized Naming Therapy: Sham tDCS plus computerized naming treatment for 15 sessions (20 minutes per each 45 minute treatment session) over the course of 3-5 weeks. Current will be administered in the in a ramp like fashion for 15-30 seconds but then the current is gradually decreased and drop to 0 mA. Language therapy will be a computer delivered naming +picture matching task.
  Sham: 2 mA of Anodal or Cathodal tDCS is induced between two 5cm X 5cm saline soaked sponges where one sponge (anode in group Anode and cathode in group Cathode) is placed on the right cerebellum. Ramping up of the current to 2 mA occurs over 15-30 seconds and then the current will be ramped back down to 0 mA in the sham condition. Termination of the stimulation after the ramping up process is generally undetectable, and the brief duration of stimulation yields no functional effects.
  Computerized naming therapy: Computer delivered naming treatment requires matching (heard and seen being produced by the speaker) with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red button if the word does not match the picture.
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 21 | 20
score on a scale | 8.31 [3.60 to 13.03] | 1.18 [-2.85 to 5.22]

3. Secondary Outcome: Change in Accuracy of Naming Untrained Pictures (Philadelphia Naming Test:PNT) Pre-treatment to 2 Months Post-treatment.
Description: as for outcome 1
Time Frame: Pre-treatment and at 2 months Post-treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 5 participants for tDCS and 3 for sham.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 21 | 21
score on a scale | 9.03 [4.31 to 13.74] | 0.38 [-3.58 to 4.36]

4. Secondary Outcome: Change in Functional Communication Skills on the ASHA-FACS Communication Independence Scale Pre-treatment to Post-treatment
Description: The American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) will be administered at Pre- treatment and Post-treatment to evaluate changes in functional communication skills.The ASHA-FACS Communication Independence scale measures functional communication performance along a continuum of independence, in terms of levels of assistance and/or prompting needed in-order to communicate. The 7-point scale ranges from 1) "does not perform the behavior" to 7) "does perform the behavior". Higher scores means better functional communication independence.
  of communication independence Scale (CI)
Time Frame: Before and after 15 sessions (3-5 sessions per week; up to 5 weeks) of treatment.
Population: Completers sample. Missing data is not imputed. The data was missing for 3 participants for tDCS and 1 participant for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 23 | 23
score on a scale | 0.27 [0.12 to 0.42] | 0.11 [-0.04 to 0.28]

5. Secondary Outcome: Change in Functional Communication Skills on the ASHA-FACS Communication Independence Scale Pre-treatment to 2 Weeks Post-treatment
Description: The American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) will be administered pre- treatment and 2 weeks post treatment to evaluate changes in functional communication skills.The ASHA-FACS Communication Independence scale measures functional communication performance along a continuum of independence, in terms of levels of assistance and/or prompting needed in-order to communicate. The 7-point scale ranges from 1) "does not perform the behavior" to 7) "does perform the behavior". Higher scores means better functional communication independence.
Time Frame: Pre-treatment and at 2 weeks Post-treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 5 participants for tDCS and 3 for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 21 | 21
score on a scale | 0.28 [0.12 to 0.44] | 0.35 [0.18 to 0.52]

6. Secondary Outcome: Change in Functional Communication Skills on the ASHA-FACS Communication Independence Scale Pre-treatment to 2 Months Post-treatment
Description: The American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) will be administered pre- treatment and 2 months post treatment to evaluate changes in functional communication skills.The ASHA-FACS Communication Independence scale measures functional communication performance along a continuum of independence, in terms of levels of assistance and/or prompting needed in-order to communicate. The 7-point scale ranges from 1) "does not perform the behavior" to 7) "does perform the behavior". Higher scores means better functional communication independence.
Time Frame: Pre-treatment and at 2 months Post-treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 6 participants for tDCS and 3 participants for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 20 | 21
score on a scale | 0.278 [0.119 to 0.436] | 0.251 [0.080 to 0.422]

7. Secondary Outcome: Change in Functional Communication Skills on the ASHA-FACS Qualitative Dimensions of Communication Scale Pre-treatment to Post-treatment
Description: The American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) will be administered pre-treatment and post-treatment to evaluate changes in functional communication skills. The ASHA-FACS Qualitative Dimensions of Communication Scale is rated on a 5-point scale reflecting adequacy, appropriateness, and promptness of communication and communication sharing.
  The 5-point scale ranges from 1) "communication is never relevant/without delay" to 5) "communication is always relevant/ without delay". Higher scores means better functional communication outcome.
Time Frame: Before and after 15 sessions (3-5 sessions per week; up to 5 weeks) of treatment.
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 23 | 23
score on a scale | 0.33 [0.20 to 0.46] | 0.04 [-0.02 to 0.11]

8. Secondary Outcome: Change in Functional Communication Skills on the ASHA-FACS Qualitative Dimensions of Communication Scale Pre-Treatment to 2 Week Post-Treatment
Description: The American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) will be administered pre-treatment and 2 weeks post-treatment to evaluate changes in functional communication skills. The ASHA-FACS Qualitative Dimensions of Communication Scale is rated on a 5-point scale reflecting adequacy, appropriateness, and promptness of communication and communication sharing. The 5-point scale ranges from 1) "communication is never relevant/without delay" to 5) "communication is always relevant/ without delay". Higher scores means better functional communication outcome.
Time Frame: Pre-treatment and at 2 weeks Post-treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 5 participants for tDCS and 3 participants for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 21 | 21
score on a scale | 0.329 [0.188 to 0.470] | 0.047 [-0.026 to 0.121]

9. Secondary Outcome: Change in Functional Communication Skills on the ASHA-FACS Qualitative Dimensions of Communication Scale Pre-treatment to 2 Months Post-treatment
Description: The American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) will be administered pre-treatment and 2 months post-treatment to evaluate changes in functional communication skills. The ASHA-FACS Qualitative Dimensions of Communication Scale is rated on a 5-point scale reflecting adequacy, appropriateness, and promptness of communication and communication sharing. The 5-point scale ranges from 1) "communication is never relevant/without delay" to 5) "communication is always relevant/ without delay". Higher scores means better functional communication outcome.
Time Frame: Pre-treatment and at 2 months Post-treatment
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 20 | 21
score on a scale | 0.351 [0.212 to 0.490] | 0.044 [-0.030 to 0.117]

10. Secondary Outcome: Change in Discourse Ability Pre-treatment to Post-treatment.
Description: The investigators will record the administration of the Cinderella Story Discourse Analysis task to compare changes in core production of words from pre-treatment to post-treatment.
  The investigators will transcribe the story told by participants at pre and post-treatment and count the total number of words produced on a Core Lexicon checklist. There are 95 words on the Core Lexicon checklist which conveys the story of Cinderella. A person earns one point for each word produced from the checklist when telling the story. Production scores range from 0-95 with higher scores associated with better performance on this discourse task.
Time Frame: Before and after 15 sessions (3-5 sessions per week; up to 5 weeks) of treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 9 participants for tDCS and 4 participants for sham.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 17 | 20
score on a scale | 1.28 [-1.43 to 3.99] | -1.03 [-4.46 to 2.40]

11. Secondary Outcome: Change in Discourse Ability Pre- Treatment to 2 Weeks Post-treatment.
Description: The investigators will record the administration of the Cinderella Story Discourse Analysis task to compare changes in core production of words from pre- treatment to 2 weeks post treatment.
  The investigators will transcribe the story told by participants at pre and post-treatment and count the total number of words produced on a Core Lexicon checklist. There are 95 words on the Core Lexicon checklist which conveys the story of Cinderella. A person earns one point for each word produced from the checklist when telling the story. Production scores range from 0-95 with higher scores associated with better performance on this discourse task.
Time Frame: Pre-treatment and at 2 weeks Post-treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 9 participants for tDCS and sham.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 17 | 15
score on a scale | 0.52 [-2.17 to 3.22] | -2.119 [-5.84 to 1.61]

12. Secondary Outcome: Change in Discourse Ability Pre-treatment to 2 Months Post-treatment.
Description: The investigators will record the administration of the Cinderella Story Discourse Analysis task to compare changes in core production of words from Pre-treatment to 2 months Post-treatment.
  The investigators will transcribe the story told by participants at pre and 2 months post-treatment and count the total number of words produced on a Core Lexicon checklist. There are 95 words on the Core Lexicon checklist which conveys the story of Cinderella. A person earns one point for each word produced from the checklist when telling the story. Production scores range from 0-95 with higher scores associated with better performance on this discourse task.
Time Frame: Pre-treatment and at 2 months Post-treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 12 participants for tDCS and 9 participants for sham
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
Number analyzed (Participants) | 14 | 15
score on a scale | 1.63 [-1.22 to 4.48] | 0.36 [-3.28 to 4.01]

ADVERSE EVENTS:
Time Frame: Up to 7 months
Groups:
- Sham Plus Computerized Naming Therapy: Sham tDCS plus computerized naming treatment for 15 sessions (20 minutes per each 45 minute treatment session) over the course of 3-5 weeks. Current will be administered in the in a ramp like fashion for 15-30 seconds but then the current is gradually decreased and drop to 0 mA. Language therapy will be a computer delivered naming +picture matching task.
  Sham: 2 mA of Anodal tDCS or Cathodal tDCS is induced between two 5cm X 5cn saline soaked sponges where one sponge (anode in group Anode and cathode in group Cathode) is placed on the right cerebellum. Ramping up of the current to 2 mA occurs over 15-30 seconds, and the current will be ramped back down to 0 mA in the sham condition. Termination of the stimulation after the ramping up process is generally undetectable, and the brief duration of stimulation yields no functional effects.
  Computerized naming therapy: Computer delivered naming treatment requires matching (heard and seen being produced by the speaker) with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red button if the word does not match the picture.
Arm/Group | tDCS Plus Computerized Naming Therapy | Sham Plus Computerized Naming Therapy
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 9/26 | 9/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS Plus Computerized Naming Therapy (N=26) | Sham Plus Computerized Naming Therapy (N=24)
Application site irritation (General disorders) | 3 (8) | 2 (2)
Application site itching (General disorders) | 6 (23) | 8 (22)
Application site burning (General disorders) | 1 (1) | 0 (0)
Application site tingling (General disorders) | 2 (7) | 2 (5)
Application site pain (General disorders) | 3 (5) | 2 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT02901574/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT02901574/ICF_000.pdf